CLINICAL TRIAL: NCT01504074
Title: Morphological and Functional Evaluation of Irvine-Gass Syndrome
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marion Munk, MD, Principal Investigator, Department of Ophthalmology and Optometry,, Medical University of Vienna
Other Study IDs: 071/2009
Record Dates: First submitted 2011-12-28; First posted 2012-01-05 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Irvine Gass Syndrome
Keywords: Irvine Gass syndrome; multimodal imaging; SD-OCT; CME secondary to cataract surgery; in vivo correlation of morphology and function
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients suffering on CME secondary to cataract surgery
  Interventions: Behavioral: if needed (decided individually) either Acular eye drops, Ultracortenol eye drop or intravitreal triamcinolone injection

INTERVENTIONS:
Behavioral: if needed (decided individually) either Acular eye drops, Ultracortenol eye drop or intravitreal triamcinolone injection — if prescribed: Ultracortenol/ Acular eye drops 3-4 times a day, if prescribed: singular intravitreal triamcinolone injection

SUMMARY:
Purpose: To evaluate morphological and functional characteristics of Irvine Gass syndrome

Methods: 30 patients suffering on Cystoid macular edema (CME) secondary to Cataract surgery will be observed and evaluated by fluorescein-angiography, SD-OCT, reading performance, contrast sensitivity and microperimetry in a fixed time schedule

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* St.p Cataract surgery
* able to read
* informed consent
* with fluorescein angiography and SD-OCT diagnosed Irvine Gass syndrome

Exclusion Criteria:

* < 18 years
* CME of other origin
* diabetic macular edema

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients suffering on CME secondary to cataract surgery
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reduction of central retinal thickness | 3 months

SECONDARY OUTCOMES:
Increase of Best corrected visual acuity | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology Medical University of Vienna, Vienna, Vienna, Austria